CLINICAL TRIAL: NCT01543802
Title: A Phase II Window-of-opportunity Study of Preoperative Therapy With Pazopanib (Votrient®) in High-risk Soft Tissue Sarcoma
Brief Title: Study of Preoperative Therapy With Pazopanib (Votrient®) to Treat High-risk Soft Tissue Sarcoma
Acronym: NOPASS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Heidelberg University (Other)
Collaborators: Universitätsmedizin Mannheim (Other); Klinikum Frankfurt Höchst (Other); German Cancer Research Center (Other); GlaxoSmithKline (Industry); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Peter Hohenberger, Head, Division of Surgical Oncology and Thoracic Surgery, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GISG-04
Record Dates: First submitted 2012-02-10; First posted 2012-03-05 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2015-12

CONDITIONS: Sarcoma, Soft-tissue
Keywords: soft-tissue sarcoma; pazopanib; antiangiogenetic treatment; endothelial progenitor cells; preoperative therapy
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental)
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — Treatment with pazopanib 800 mg qd for 21 days followed by resection of the tumor after a 7-14 days break
  Other Names: Votrient

SUMMARY:
The purpose of this study is to examine if a short-term treatment with pazopanib, an oral drug inhibiting the growth of blood vessel, can reduce the metabolism of soft-tissue sarcomas and thus facilitate their resection when given prior to surgery. Moreover, the study assesses the prognostic and predictive value of several new biomarkers (endothelial progenitor cells, soluble vascular epithelial growth factor),

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.
2. Age ≥ 18 years or legal age of consent if different from 18 years.
3. Non-metastatic primary tumor or locoregional recurrence of histologically confirmed high-risk (G2/3, diameter ≥5 cm) soft tissue sarcoma (STS) of any location (extremities, girdle, trunk, retroperitoneum); or metachronous solitary metastasis of STS for which surgical resection is planned according to the individual choice of the multidisciplinary treatment team (no grade or size restrictions apply for metastasis).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Measurable disease according to RECIST 1.1
6. Resectable and solitary tumor, as assessed by the investigator based on staging exams (CT scan of the chest, CT or MRI of the abdomen, MRI of the limb in case of extremity STS).
7. Adequate organ system function
8. Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of study treatment and agree to use effective contraception, during the study and until after surgery has been performed.
9. Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

1. The following tumor types are ineligible

   * Embryonal rhabdomyosarcoma
   * Chondrosarcoma
   * Osteosarcoma
   * Ewing tumors / PNET
   * Gastro-intestinal stromal tumors
   * Dermofibromatosis sarcoma protuberans
   * Inflammatory myofibroblastic sarcoma
   * Malignant mesothelioma
2. Prior malignancy.
3. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis.
4. Prior or concurrent systemic chemotherapy or molecularly targeted therapy for STS or other malignancies within five years before study entry.
5. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
6. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
7. Corrected QT interval (QTc) > 480 msecs (calculation according to Bazett).
8. Presence of uncontrolled infection.
9. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
10. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].
11. Cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
12. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement are not considered to be major surgery).
13. Evidence of active bleeding or bleeding diathesis.
14. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
15. Recent hemoptysis (more than ½ teaspoon of red blood within 8 weeks before first dose of study drug).
16. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
17. Inability or unwillingness to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of investigational product and for the duration of the study.
18. Treatment with any of the following therapies:

    * radiation therapy, surgery targeting the lesion under study other than incisional biopsy, or tumor embolization, prior to the first dose of pazopanib OR
    * chemotherapy, immunotherapy, biologic therapy, antiangiogenic therapy, investigational therapy or hormonal therapy, targeting the lesion under study, prior to the first dose of pazopanib OR
    * chemotherapy, immunotherapy, biologic therapy, antiangiogenic therapy, investigational therapy or hormonal therapy, targeting any other lesion / disease, within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib
19. Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment.
20. Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity, except alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Metabolic response rate | day 22-28 (time of post-treatment PET-CT)
  Metabolic response rate is defined as the proportion of patients achieving a metabolic response, i.e. a 50% reduction of the mean standardized uptake value (SUVmean) in the post-treatment compared to the pre-treatment FDG-PET-CT

SECONDARY OUTCOMES:
Percentage of tumor tissue with regressive alterations upon resection ("Histopathological Response") | day 28-35
Decrease in tumor size in MRI according to RECIST 1.1 criteria | baseline and day 22-28
Change of FDG influx as well as of transport rates k1-k4 and distribution volume VB and fractal dimension in dynamic PET-CT ("Dynamic PET-CT Response") | baseline and day 22-28
  Absolute values of all parameters of FDG kinetics will be used for discriminant analysis evaluation.
Number of days for which planned resection is delayed after treatment | day 28-35
Number of patients in which adverse events occur during treatment | day 1-21
  Adverse events are graded according to NCI Common Terminology Criteria for Adverse Events v4.0 (NCI CTCAE v4)
Disease-free survival | 3 years
Local recurrence-free survival | 3 years
Distant recurrence-free survival | 3 years
Overall survival | 3 years
Decrease in vascularisation in MRI according to adapted Choi Criteria | baseline and day 22-28
  Adapted Choi Criteria as defined ín Stacchiotti S, Collini P, Messina A, Morosi C, Barisella M, Bertulli R, et al. High-grade soft-tissue sarcomas: tumor response assessment--pilot study to assess the correlation between radiologic and pathologic response by using RECIST and Choi criteria. Radiology 2009;251(2):447-56.
Decrease in MRI apparent diffusion coefficient (ADC) values | baseline and day 22-28
  ADC values as defined by Dudeck O, Zeile M, Pink D, Pech M, Tunn PU, Reichardt P, et al. Diffusion-weighted magnetic resonance imaging allows monitoring of anticancer treatment effects in patients with soft-tissue sarcomas. J Magn Reson Imaging 2008;27(5):1109-13.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hohenberger, MD, Principal Investigator — University Hospital Mannheim, Department of Surgery
Locations (4):
- Germany (4):
  - Klinikum Frankfurt-Höchst, Frankfurt am Main
  - German Cancer Research Center, Medical PET Group - Biological Imaging, Heidelberg
  - University Hospital Heidelberg / National Centre for Tumor Diseases, Heidelberg
  - University Hospital Mannheim, Dpt. of Surgery, Mannheim

REFERENCES:
- [Derived] Ronellenfitsch U, Karampinis I, Dimitrakopoulou-Strauss A, Sachpekidis C, Jakob J, Kasper B, Nowak K, Pilz L, Attenberger U, Gaiser T, Derigs HG, Schwarzbach M, Hohenberger P. Preoperative Pazopanib in High-Risk Soft Tissue Sarcoma: Phase II Window-of Opportunity Study of the German Interdisciplinary Sarcoma Group (NOPASS/GISG-04). Ann Surg Oncol. 2019 May;26(5):1332-1339. doi: 10.1245/s10434-019-07183-4. Epub 2019 Mar 6. PMID 30843160
- [Derived] Ronellenfitsch U, Dimitrakopoulou-Strauss A, Jakob J, Kasper B, Nowak K, Pilz LR, Attenberger U, Gaiser T, Egerer G, Frohling S, Derigs HG, Schwarzbach M, Hohenberger P. Preoperative therapy with pazopanib in high-risk soft tissue sarcoma: a phase II window-of-opportunity study by the German Interdisciplinary Sarcoma Group (GISG-04/NOPASS). BMJ Open. 2016 Jan 6;6(1):e009558. doi: 10.1136/bmjopen-2015-009558. PMID 26739732
- See also: General info on German Interdisciplinary Sarcoma Group, under whose auspices the trial is conducted — http://www.gisg.de